CLINICAL TRIAL: NCT06870396
Title: National Study of Adrenal Tumours
Acronym: NSAT
Status: Enrolling by invitation | Type: Observational
Sponsor: Society for Endocrinology (Other)
Responsible Party: Sponsor
Other Study IDs: NSAT2024.01
Record Dates: First submitted 2024-11-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pheochromocytoma and Paraganglioma (PPGL); Adrenocorticol Cancer (ACC); Adrenal Tumours
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a study putting together large numbers of patients with or without a hereditary risk of adrenal tumours including tumours such as adrenocortical carcinoma and phaeochromocytoma/paraganglioma. The purpose is to answer questions about the survival of patients with these rare tumours and to do this, we will collect information on diagnosis and management of these tumours. This data will be best assessed by combing these rare cases at a national level recruiting from centres throughout UK and Ireland. The information will be confidential and stored in a secure platform.

Patients will be approached for consent to gather their data by their local consultants and patients will have the choice to participate or decline participation, which will not affect their standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of phaeochromocytoma or paraganglioma or adrenocortical tumour based on histology and or biochemical testing including plasma or urine metanephrine's or a urine steroid profile and confirmatory imaging tests or patients with a confirmed pathogenic variant in a known PPGL predisposition gene
2. Patient is willing and able to give informed consent for the participation in the study.
3. Male or female, and over the age of 18.
4. Patient, in the investigator's opinion, is able and willing to comply with all the study requirements.
5. Patients held on local hospital audit notes who have had a diagnosis of phaeochromocytoma or paraganglioma or adrenocortical tumour based on histology and or biochemical testing including plasma or urine metanephrine's or a urine steroid profile and confirmatory imaging tests or patients with a confirmed pathogenic variant in a known PPGL predisposition gene who are now deceased and have been deceased prior to the start of the study.

Exclusion Criteria:

1. Alive patients unable to give informed consent will not be recruited
2. Patients with an unconfirmed diagnosis of phaeochromocytoma or paraganglioma or adrenocortical tumour based on histology and or biochemical testing including plasma or urine metanephrine's or a urine steroid profile and confirmatory imaging tests or patients with unconfirmed pathogenic variant in a known PPGL predisposition gene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of phaeochromocytoma or paraganglioma or adrenocortical tumour based on histology and or biochemical testing including plasma or urine metanephrine's or a urine steroid profile and confirmatory imaging tests or patients with a confirmed pathogenic variant in a known PPGL predisposition gene
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2034-06-30 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
review outcome data and calculate median overall survival for patients with metastatic pheochromocytoma and paraganglioma (PPGL) and adrenocortical carcinoma (ACC) using existing standard of are therapies over the past 10 years | 10 years
  Primary aims:
  i) identify the clinical need within the UK, ii) review outcome data and calculate median overall survival for patients with metastatic pheochromocytoma and paraganglioma (PPGL) and adrenocortical carcinoma (ACC) using existing standard of care therapies over the past 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge NHS, Cambridge, UK, United Kingdom